CLINICAL TRIAL: NCT04039672
Title: Interest of Tumor Replicates in Avian Embryo to Model Therapeutic Effects of BRAF Inhibitors/MEK Inhibitors (BRAFi/MEKi) in BRAF Mutated Melanoma
Brief Title: Interest of Tumor Replicates in Avian Embryo to Model Therapeutic Effects of BRAFi/MEKi in BRAF Mutated Melanoma
Acronym: MELANOPREDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL19_0248
Record Dates: First submitted 2019-05-15; First posted 2019-07-31 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Melanoma
Keywords: Melanoma; Avian embryo
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biopsy (Experimental): Skin biopsy before BRAFi/MEKi treatment
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Procedure: Skin biopsy — 5mm skin metastasis or primary melanoma biopsy

SUMMARY:
This is an interventional mono-centric study in patients with BRAF mutated metastatic melanoma treated with BRAF/MEK inhibitors. The aim of the study is to test the grafting of patient tumoral cells in avian embryo and develop a predictive in vivo model for patient treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Signed written informed consent
* Patient with BRAF V600 mutated metastatic or unresectable melanoma histologically confirmed
* BRAFi/MEKi treatment indication
* Patient with skin tumor (excluded face and skinfold) available for biopsy
* Measurable disease as defined by RECIST v1.1 criteria
* Patient affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Ocular melanoma
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
* Pregnant or nursing (lactating) women
* Patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Grafted avian embryo development | 2 days post graft
  Number of grafted embryo which develop tumor measurable by 3D microscopy
Grafted avian embryo viability | 2 days post graft
  Survival rate of grafted embryo

SECONDARY OUTCOMES:
BRAFi/MEKi maximum toxic effect dose in avian embryo | 3 months post treatment administration
  Survival rate in avian embryo after treatment injections in different concentrations
BRAFi maximum toxic effect dose in avian embryon | 3 months post treatment administration
  Survival rate in avian embryo after treatment injections in different concentrations
MEKi maximum toxic effect dose in avian embryo | 3 months post treatment administration
  weight of avian embryo after treatment injections in different concentrations
BRAFi maximum toxic effect dose in avian embryo | 3 months post treatment administration
  Height of avian embryo after treatment injections in different concentrations
MEKi maximum toxic effect dose in avian embryo | 3 months post treatment administration
  Height of avian embryo after treatment injections in different concentrations
BRAFi maximum toxic effect dose in avian embryo | 3 months post treatment administration
  Presence of cardiac malformation in avian embryo after treatment injections in different concentrations
MEKi maximum toxic effect dose in avian embryo | 3 months post treatment administration
  Presence of cardiac malformation in avian embryo after treatment injections in different concentrations
BRAFi maximum toxic effect dose in avian embryo | 3 months post treatment administration
  Presence of craniofacial malformation in avian embryo after treatment injections in different concentrations
MEKi maximum toxic effect dose in avian embryo | 3 months post treatment administration
  Presence of craniofacial malformation in avian embryo after treatment injections in different concentrations
Patient treatment response | 3 months post inclusion
  RECIST 1.1 response
Embryo treatment response (tumor) | 2 days post graft
  Embryo tumor volume obtained by confocal microscopy before treatment administration compared with tumor volume of non-treated embryo
Embryo treatment response (metastasis) | 2 days post graft
  Metastasis appearance

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Dermatologie, Centre hospitalier Lyon Sud, HCL, Pierre-Bénite, France